CLINICAL TRIAL: NCT01394757
Title: Brain Network Dysfunction as a Model for Schizophrenia: Connectivity Alterations Using Ketamine and Pharmacological Magnetic Resonance Imaging
Brief Title: Network Dysfunction, Schizophrenia and Pharmacological Magnetic Resonance Imaging (phMRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: P14193ONB; 2010-022772-31 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Esketamine hydrochloride — Bolus: 15 mg/kg over 1 minute, followed by a maintenance infusion of 0.25 mg/kg/h for 19 minutes.
  Other Names: Ketanest S; Ketamine

SUMMARY:
Alterations of functional brain networks have been frequently demonstrated in schizophrenia, although the exact underlying molecular mechanisms remain unrevealed. Ketamine is known to exert its schizophrenia-like effects through modulation of the glutamatergic system, thus facilitating the investigation of the impact of this specific transmitter system on resting state functional brain networks. The aim of the study is therefore to use pharmacological functional Magnetic Resonance Imaging (phMRI) to examine changes in brain networks involved in schizophrenia in response to ketamine application compared to placebo. 30 healthy subjects (15 females) will be examined twice using a double-blind, placebo-controlled, randomized, crossover, counterbalanced-order design. Resting state fMRI will be investigated before, during and after either placebo or ketamine intravenous infusion for 20 minutes. Prior to the main trial 10 additional participants will be included in an open pilot trial.

Hypothesis: Ketamine application will induce changes in resting state networks previously associated with schizophrenia and in the connectivity of relevant brain regions such as the striatum, thalamus, caudate, hippocampus and amygdala. Furthermore, the application of ketamine will provoke changes in the BOLD-activation in three fMRI paradigms each performed before and after ketamine infusion.

ELIGIBILITY:
Inclusion Criteria:

* general health based on history, physical examination, ECG, laboratory screening and structured clinical interview for DSM-IV(SCID)
* willingness and competence to sign the informed consent form
* aged 18 to 55 years

Exclusion Criteria:

* any medical, psychiatric or neurological illness
* current or former substance abuse
* any implant or stainless steel graft and any other contraindications for MRI
* pregnancy
* first degree relatives with a history of psychiatric illness or substance abuse
* failures to comply with the study protocol or to follow the instructions of the investigating team
* lifetime use of antipsychotic drugs
* treatment with psychotropic agents such as SSRIs within the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Ketamine-induced changes in BOLD-activity over time | 1 year
  participants will be measured twice and all participants are expected to be recruited and measured within 1 year

SECONDARY OUTCOMES:
Change of task-induced BOLD-activity by ketamine application | 60 minutes (before and after ketamine infusion) at each MRI session (interval between MRI scans: 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, A/Prof., MD, Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- See also: Homepage of the Functional Neuroimaging Group, Department of Psychiatry and Psychotherapy, Medical University of Vienna — http://www.meduniwien.ac.at/neuroimaging/